CLINICAL TRIAL: NCT06312072
Title: Understanding Risk Factors for Progressive Chronic Kidney Disease in Malawi to Inform Interventions for Earlier Detection and Prevention (Impso Study)
Brief Title: Understanding Risk Factors for Progressive Chronic Kidney Disease in Malawi
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Wellcome Trust (Other); Malawi Epidemiology and Intervention Research Unit (Other); London School of Hygiene and Tropical Medicine (Other); University of Glasgow (Other); Malawi-Liverpool-Wellcome Trust Clinical Research Programme (Other)
Responsible Party: Sponsor
Other Study IDs: 23-019
Record Dates: First submitted 2023-04-11; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2023-04

CONDITIONS: Chronic Kidney Diseases; Non-Communicable Chronic Diseases; Non-communicable Disease; Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic; Noncommunicable Diseases; Kidney Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Serum (blood) samples will be stored in MEIRU's biorepository for use in future longitudinal studies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MEIRU rural population cohort: Adults aged >=18 living in MEIRU's rural health demographic surveillance area (Karonga district)
  No interventions to be administered; observational study only, with collection of survey data, blood samples and urine samples.
  Interventions: Other: No intervention; observational study
- MEIRU urban population cohort: Adults aged >=18 living in MEIRU's urben demographic surveillance area (Lilongwe Area 25)
  No interventions to be administered; observational study only, with collection of survey data, blood samples and urine samples.
  Interventions: Other: No intervention; observational study

INTERVENTIONS:
Other: No intervention; observational study — No intervention; observational study

SUMMARY:
Worldwide, the number of people living with long-term health conditions, including chronic kidney disease (CKD), is increasing. CKD is usually asymptomatic in early stages but can progress to advanced disease, including kidney failure, causing significant morbidity and mortality.

In low-income countries of sub-Saharan Africa, including Malawi, treatments for kidney failure are not yet widely available and are prohibitively expensive . It is therefore vital to:

(a) Prevent development of CKD in the first place (b) Detect CKD earlier so that more cost-effective treatments can be given to slow progression.

There is little evidence on factors that drive CKD progression in Malawi, or on interventions that may be cost-effective for improving detection and slowing disease progression in this setting. This PhD will address these knowledge gaps, through the following aims:

1) Determine the mortality associated with CKD, and the risk factors driving its development and progression in Malawian adults 2) Investigate the impacts of different models for integrating screening and prevention strategies for CKD and its risk factors into health services for other long-term conditions in low- and middle-income countries 3) With patients, carers, healthcare workers and policy makers, evaluate the feasibility and acceptability of different potential models for integrating CKD screening and prevention strategies into health services for high-risk patient groups in Malawi

DETAILED DESCRIPTION:
Background:

CKD prevalence is rising most rapidly in sub-Saharan Africa (current estimates 13-15%), where health systems are least equipped to tackle it (1-7). Malawi has only one nephrologist for a population of over 19 million and kidney replacement therapy (KRT), which consumes disproportionate healthcare spending, remains extremely limited (8,9).

Historically there has been insufficient data on CKD in LMICs owing to difficulties accessing diagnostics and uncertainty regarding the most appropriate context-specific methods for estimating kidney function (10).

Recent research by the African Research on Kidney Disease (ARK) group using measured GFR has shown that previous creatinine-based estimates significantly underestimated CKD burden in many African countries; in Malawi prevalence of eGFR <90ml/min/1.73m2 may be 51%, and eGFR <60ml/min/1.73m2 as high as 11.9% (6).

CKD has many causes, impacting on the public health strategies required to tackle it; however data on its underlying causes in Malawi and other countries of low-income Africa remain limited.

Cross-sectional data suggests risk is greater in older people with other LTCs (e.g. hypertension, HIV), however other causes are unaccounted for (11-14). No longitudinal research has been conducted in Malawi to explore the impact of traditional and non-traditional risk factors on CKD development and progression.

Evidence on proteinuria in Malawi is also sparse, a well-recognised predictor for progressive kidney disease, cardiovascular morbidity and mortality (15-17) and a therapeutic target of drugs mitigating progression (18-22).

Early detection and prevention of CKD and its risk factors, integrated with other LTCs, is vital to cost-effectively improve health outcomes within available resources, as recognised by the Malawi government's National Action Plan for NCDs (23-25). To guide this, more research is urgently needed on the risk factors for CKD development and progression in this setting, and on strategies for early detection and prevention and that may be effectively integrated with public health plans for other LTCs, without reliance on specialist nephrology input.

Aims and Objectives:

The overall work package has three main aims:

Aim 1: Determine (a) the mortality associated with CKD, and (b) the risk factors driving its development and progression in Malawian adults

Aim 2: Investigate the impacts of different models for integrating screening and prevention strategies for CKD and its risk factors into health services for other LTCs in LMICs.

Aim 3: With different stakeholder groups, qualitatively evaluate the feasibility and acceptability of different potential models for integrating CKD screening and prevention strategies into health services for high-risk patient groups in Malawi

The work described here relates to observational research which aims to address Aim 1. The specific objectives within Aim 1 are as follows:

Aim 1, Objective 1:

In Malawian adults aged ≥18 years living in MEIRU's rural +/- urban population cohorts, investigate the association between baseline kidney function and mortality outcomes (all-cause and cause-specific)

Aim 1, Objective 2:

In adults aged ≥18 years living in MEIRU's rural and urban population cohorts, determine the risk factors associated with development of impaired kidney function

Aim 1, Objective 3:

In adults aged ≥18 years living in MEIRU's rural and urban population cohorts, determine the risk factors associated with progression of impaired kidney function

Planned methods for Aim 1:

The proposed work for Aim 1 is nested within MEIRU rural (Karonga HDSS) and urban (Area 25, Lilongwe) open, population-based cohorts. These nationally representative cohort populations (n>50,000 adults ≥15 years) are situated in 135km2 of rural subsistence farming and fishing communities in northern Malawi and a township in the capital city. Population surveillance already includes annual censuses; births, deaths and migration registration, sociodemographic data and HIV-testing. This is ongoing in the rural cohort since 2002 and commenced in the urban cohort in 2022.26 For all deaths, a standardised WHO verbal autopsy (VA) tool is used to assign cause of death.

In both settings a comprehensive NCD survey was conducted 2013-2016. The currently ongoing Healthy Lives Malawi (HLM) survey is re-surveying long-term conditions (LTCs) in these populations. Available data from these two surveys includes household (SES, geolocators), interview (demographics, lifestyle factors, clinical history (prior diagnosis, screening and medications for chronic conditions), examination and measures (anthropometry, blood pressure, hand grip strength, peripheral arterial measures) and biological sample collection (serum, plasma and whole blood samples stored at -80 Celsius and other biological material).

Aim 1, objective 1

* Investigate the association between baseline kidney function and mortality outcomes (all-cause and cause-specific) in Malawian adults Study design
* Survival analysis using secondary data Study population
* Adults aged ≥18 years living within the demographic surveillance areas (Karonga HDSS +/- area 25, Lilongwe depending on availability of longitudinal data for the urban site), who participated in the 2013-16 NCD survey Approach and methods
* eGFRcreat and eGFRcystC will be calculated for adults living in the rural (+/- urban) site who have had serum creatinine (estimated n≥5000) +/- cystatin C (estimated n≥2500) tested on historical serum samples collected during their participation in the 2013-16 NCD survey, and for whom longitudinal demographic surveillance data is available
* Existing sociodemographic and comorbidity data will be available for these individuals
* Existing mortality data (physician assigned cause of death from verbal autopsy reports) will be analysed to for adults in different baseline eGFR categories
* Participants will be included until last point of follow-up

Aim 1, objective 2 - Investigate the risk factors for development of impaired kidney function in Malawian adults

Study design

* Retrospective cohort study Study population
* Adults aged ≥18 years living within the demographic surveillance areas (Karonga HDSS +/- area 25, Lilongwe), who had had eGFRcreat ≥60ml/min/1.73m2 during their participation in the 2013-16 NCD survey, and who have also participated in the follow-up 2022-25 LTC survey Approach and methods

  * A sample of n=~4000 adults with eGFRcreat ≥60ml/min/1.73m2 at baseline (2013-16) will be randomly selected within age and sex strata (these creatinine results are already available from which eGFR can be calculated)
  * The participants will have already participated in the 2022-25 LTC survey; serum and plasma samples are collected for storage in this survey and participants provide consent for testing of these samples in future studies
  * Creatinine will be tested on the 2022-25 LTC serum samples such that each participant has individual-level paired creatinine results from the two surveys
* Extensive sociodemographic and comorbidity data from both surveys already exists for all participants. These will be used to analyse associations between risk factors of interest and development of kidney disease outcome measures

Aim 1, Objective 3

* Investigate the risk factors for progression of impaired kidney function in Malawian adults Study design
* Prospective cohort study

Study population

- Adults aged ≥18 years living within the demographic surveillance areas (Karonga HDSS +/- area 25, Lilongwe), with persistent eGFRcystC <90ml/min/1.73m2 during their participation in both the 2013-16 NCD and 2022-25 LTC surveys

Approach and methods

An age-, sex- and site-stratified sample of n=1000-1100 adults with eGFRcystC <90ml/min/1.73m2 at baseline (2013-16) will be selected (serum creatinine results will also be available for these individuals)

The participants will have already participated the 2022-25 LTC survey; serum and plasma samples are collected for storage in this survey and participants provide consent for testing of these in related and future studies.

Cystatin C and creatinine will be tested on the 2022-25 LTC serum samples such that each participant has individual-level paired kidney function results from the two previous surveys.

At ≥90 days following the LTC sample collection, a medical fieldworker will visit the household of each eligible participant to invite participation and consent (or assent) to participate in data collection for kidney disease and its risk factors, using standardised procedures for recording, collecting measurements and coding.

The data collected on kidney disease and its risk factors will include:

1. A medical interview, containing questions on potential risk factors for kidney disease not already captured in the LTC survey (specific medical history, specific medications, family history)
2. Health-related quality of life data
3. HIV rapid test and counselling will be offered to individuals with unknown HIV status
4. Venepuncture for blood tests - creatinine and cystatin C (taken ≥90 days after LTC sample, confirming chronicity) and for storage
5. Early morning mid-stream urine (MSU) collection - for point of care dipstick urinalysis, and laboratory tests, including microscopy, gram stain, filtration and centrifugation (for Schistosoma ova) and urine albumin-creatinine ratio (uACR).

The medical interview and health-related quality of life questionnaire data will be collected at the first household visit following the patient information and consent process; blood and urine samples will then be collected at a second, early morning household visit. Screening questions about menstruation (for females) and symptoms of urinary tract infection will be asked prior to scheduling the second household visit. Participants with symptoms of urine infection will be referred for clinical assessment. Participants with new urine symptoms or with particular urine dipstick abnormalities (leucocytes, nitrites and/or blood) at the point of urine collection at the second household visit will receive a third household visit for collection of a second, confirmatory urine sample.

Schistosoma IgG ELISA and CRP, new risk factors of interest, will be tested on participants' stored serum samples (from 2013-16).

Data on these new risk factors of interest will be analysed for association with kidney disease progression outcomes.

ELIGIBILITY:
Aim 1, Objective 1 (survival analysis):

Inclusion Criteria:

* Adult ≥ 18 years at time of participation in 2013-16 NCD survey
* Living in one of the demographic surveillance sites (Chilumba, Karonga or Lilongwe area 25)
* Creatinine +/- cystatin C result available from serum sample taken in 2013-16 NCD survey

Exclusion Criteria:

* Child (age <18 years)
* Not living in one of the study areas

Aim 1, Objective 2 (retrospective cohort study)

Inclusion criteria:

* eGFRcreat ≥60ml/min/1.73m3 at baseline (using creatinine tested on serum sample from 2013-16 survey)
* Participated and provided blood (serum) sample in 2022-25 long-term conditions (LTC) survey i.e. individual-level longitudinal paired serum samples available, including consent already given for testing of stored samples in future studies

Exclusion Criteria:

* Child (age <18 years)
* Not living in one of the study areas
* Not consented previously to storage of blood samples and use of samples in future studies

Aim 1, Objective 3

Inclusion criteria:

As for Objective 1, PLUS:

* eGFRcystC <90ml/min/1.73m3 at baseline (using cystatin C tested on 2013-16 serum sample)
* Participated and provided serum sample in 2022-25 long-term conditions (LTC) survey i.e. individual-level longitudinal paired serum samples available
* Still alive and living in one of the demographic surveillance sites
* Able to provide consent or assent with consent from an appropriate nominated guardian

Exlusion criteria:

* Declines consent
* Unable to consent or assent
* Children (<18 years)
* Non-resident in study areas
* Acute physical or mental illness
* Hospital inpatient
* Hospital admission >24 hours in past 90 days and <90 days until study end
* Currently pregnant

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The proposed work for Aim 1 is nested within MEIRU rural (Karonga HDSS) and urban (Area 25, Lilongwe) open, population-based cohorts. These nationally representative cohort populations are situated in 135km2 of rural subsistence farming and fishing communities in northern Malawi and a township in the capital city. Population surveillance already includes annual censuses; births, deaths and migration registration, sociodemographic data and HIV-testing. This is ongoing in the rural cohort since 2002 and commenced in the urban cohort in 2022 (26). Detailed sociodemographic and risk factor data is available from two surveys (2013-16 non-communicable disease survey and 2022-25 long-term conditions survey).
Sampling Method: Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Aim 1, objective 3 primary outcome measure | Over duration of follow-up (2013 to 2025, average around 7.5 years)
  25% reduction in eGFRcystC from baseline AND change in eGFRcystC category
Aim 1, objective 2 primary outome measure | Over duration of follow-up (2013 to 2025, average around 7.5 years)
  Development of eGFRcreat <60ml/min/1.72m2
Aim 1, objective 1 primary outcome measure: | Deaths reported over maximum 10 year time period (time of inclusion in NCD study, 2013-16, to time of analysis, 2023)
  • All-cause mortality rate per 1000 person-years at risk (adjusted for age, sex, key comorbidities)

SECONDARY OUTCOMES:
Aim 1, objective 3 secondary outcome measure 1: | Over duration of follow-up (2013 to 2025, average around 7.5 years)
  25% reduction in eGFRcreat from baseline AND change in eGFRcreat category
Aim 1, objective 3 secondary outcome measure 2: | Over duration of follow-up (2013 to 2025, average around 7.5 years)
  57% decline in eGFR
Aim 1, objective 3 secondary outcome measure 3: | Over duration of follow-up (2013 to 2025, average around 7.5 years)
  40% decline in eGFR
Aim 1, objective 3 secondary outcome measure 4: | Over duration of follow-up (2013 to 2025, average around 7.5 years)
  30% decline in eGFR
Aim 1, objective 3 secondary outcome measure 5: | Over duration of follow-up (2013 to 2025, average around 7.5 years)
  20% decline in eGFR
Aim 1, objective 3 secondary outcome measure 6: | Over duration of follow-up (2013 to 2025, average around 7.5 years)
  Kidney failure, defined by:
  * eGFR<15ml/min/1.73m2
  * Commencement of maintenance KRT (≥4 weeks duration)
Aim 1, objective 2 secondary outcome measure: | Over duration of follow-up (2013 to 2025, average around 7.5 years)
  Development of eGFRcreat <90ml/min/1.72m2
Aim 1, objective 1 secondary outcome measure: | Deaths reported over maximum 10 year time period (time of inclusion in NCD study, 2013-16, to time of analysis, 2023)
  Cause-specific mortality per 1000 person-years at risk (physician-assigned)

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Snead, BM BCh, Principal Investigator — Liverpool School of Tropical Medicine
Locations (1):
- Malawi Epidemiology and Intervention Research Unit, Chilumba, Karonga, Malawi

IPD SHARING:
Plan to Share IPD: Yes
This study will contribute data to the MEIRU data repository. MEIRU has a data access management committee which will approve any requested access to MEIRU data repository.
Time Frame: The MEIRU data access management committee is responsible for deciding on data to be made publicly available, and time frames.
Access Criteria: The MEIRU data access management committee is responsible for deciding on data to be made publicly available, and time frames. Additionally, through a systematised data access requests, the committee will authorize access to more highly resolved data sets. The Biorepository Access Management Committee will approve sample access plans.

REFERENCES:
- [Background] GBD Chronic Kidney Disease Collaboration. Global, regional, and national burden of chronic kidney disease, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2020 Feb 29;395(10225):709-733. doi: 10.1016/S0140-6736(20)30045-3. Epub 2020 Feb 13. PMID 32061315
- [Background] Eckardt KU, Coresh J, Devuyst O, Johnson RJ, Kottgen A, Levey AS, Levin A. Evolving importance of kidney disease: from subspecialty to global health burden. Lancet. 2013 Jul 13;382(9887):158-69. doi: 10.1016/S0140-6736(13)60439-0. Epub 2013 May 31. PMID 23727165
- [Background] Levin A, Tonelli M, Bonventre J, Coresh J, Donner JA, Fogo AB, Fox CS, Gansevoort RT, Heerspink HJL, Jardine M, Kasiske B, Kottgen A, Kretzler M, Levey AS, Luyckx VA, Mehta R, Moe O, Obrador G, Pannu N, Parikh CR, Perkovic V, Pollock C, Stenvinkel P, Tuttle KR, Wheeler DC, Eckardt KU; ISN Global Kidney Health Summit participants. Global kidney health 2017 and beyond: a roadmap for closing gaps in care, research, and policy. Lancet. 2017 Oct 21;390(10105):1888-1917. doi: 10.1016/S0140-6736(17)30788-2. Epub 2017 Apr 20. PMID 28434650
- [Background] Stanifer JW, Jing B, Tolan S, Helmke N, Mukerjee R, Naicker S, Patel U. The epidemiology of chronic kidney disease in sub-Saharan Africa: a systematic review and meta-analysis. Lancet Glob Health. 2014 Mar;2(3):e174-81. doi: 10.1016/S2214-109X(14)70002-6. Epub 2014 Feb 10. PMID 25102850
- [Background] Kaze AD, Ilori T, Jaar BG, Echouffo-Tcheugui JB. Burden of chronic kidney disease on the African continent: a systematic review and meta-analysis. BMC Nephrol. 2018 Jun 1;19(1):125. doi: 10.1186/s12882-018-0930-5. PMID 29859046
- [Background] Fabian J, Kalyesubula R, Mkandawire J, Hansen CH, Nitsch D, Musenge E, Nakanga WP, Prynn JE, Dreyer G, Snyman T, Ssebunnya B, Ramsay M, Smeeth L, Tollman S, Naicker S, Crampin A, Newton R, George JA, Tomlinson L; African Research on Kidney Disease Consortium. Measurement of kidney function in Malawi, South Africa, and Uganda: a multicentre cohort study. Lancet Glob Health. 2022 Aug;10(8):e1159-e1169. doi: 10.1016/S2214-109X(22)00239-X. PMID 35839814
- [Background] Luyckx VA, Moosa MR. Priority Setting as an Ethical Imperative in Managing Global Dialysis Access and Improving Kidney Care. Semin Nephrol. 2021 May;41(3):230-241. doi: 10.1016/j.semnephrol.2021.05.004. PMID 34330363
- [Background] Dreyer G, Dobbie H, Banks R, Allain T, Gonani A, Turner NLV. Supporting Malawi's dialysis services in the international community. Br J Ren Med. 2012;17:24-6.
- [Background] https://www.theisn.org/blog/2014/11/24/caring-for-kidney-patients-in-malawi/
- [Background] Fabian J, George JA, Etheredge HR, van Deventer M, Kalyesubula R, Wade AN, Tomlinson LA, Tollman S, Naicker S. Methods and reporting of kidney function: a systematic review of studies from sub-Saharan Africa. Clin Kidney J. 2019 Aug 19;12(6):778-787. doi: 10.1093/ckj/sfz089. eCollection 2019 Dec. PMID 31807291
- [Background] Nakanga WP, Prynn JE, Banda L, Kalyesubula R, Tomlinson LA, Nyirenda M, Crampin AC. Prevalence of impaired renal function among rural and urban populations: findings of a cross-sectional study in Malawi. Wellcome Open Res. 2019 Jun 10;4:92. doi: 10.12688/wellcomeopenres.15255.1. eCollection 2019. PMID 31656860
- [Background] Muiru AN, Charlebois ED, Balzer LB, Kwarisiima D, Elly A, Black D, Okiror S, Kabami J, Atukunda M, Snyman K, Petersen M, Kamya M, Havlir D, Estrella MM, Hsu CY. The epidemiology of chronic kidney disease (CKD) in rural East Africa: A population-based study. PLoS One. 2020 Mar 4;15(3):e0229649. doi: 10.1371/journal.pone.0229649. eCollection 2020. PMID 32130245
- [Background] Kalyesubula R, Nankabirwa JI, Ssinabulya I, Siddharthan T, Kayima J, Nakibuuka J, Salata RA, Mondo C, Kamya MR, Hricik D. Kidney disease in Uganda: a community based study. BMC Nephrol. 2017 Apr 3;18(1):116. doi: 10.1186/s12882-017-0521-x. PMID 28372551
- [Background] Stanifer JW, Maro V, Egger J, Karia F, Thielman N, Turner EL, Shimbi D, Kilaweh H, Matemu O, Patel UD. The epidemiology of chronic kidney disease in Northern Tanzania: a population-based survey. PLoS One. 2015 Apr 17;10(4):e0124506. doi: 10.1371/journal.pone.0124506. eCollection 2015. PMID 25886472
- [Background] Ruggenenti P, Perna A, Mosconi L, Matalone M, Pisoni R, Gaspari F, Remuzzi G. Proteinuria predicts end-stage renal failure in non-diabetic chronic nephropathies. The "Gruppo Italiano di Studi Epidemiologici in Nefrologia" (GISEN). Kidney Int Suppl. 1997 Dec;63:S54-7. PMID 9407422
- [Background] Peterson JC, Adler S, Burkart JM, Greene T, Hebert LA, Hunsicker LG, King AJ, Klahr S, Massry SG, Seifter JL. Blood pressure control, proteinuria, and the progression of renal disease. The Modification of Diet in Renal Disease Study. Ann Intern Med. 1995 Nov 15;123(10):754-62. doi: 10.7326/0003-4819-123-10-199511150-00003. PMID 7574193
- [Background] Agrawal V, Marinescu V, Agarwal M, McCullough PA. Cardiovascular implications of proteinuria: an indicator of chronic kidney disease. Nat Rev Cardiol. 2009 Apr;6(4):301-11. doi: 10.1038/nrcardio.2009.11. PMID 19352334
- [Background] Randomised placebo-controlled trial of lisinopril in normotensive patients with insulin-dependent diabetes and normoalbuminuria or microalbuminuria. The EUCLID Study Group. Lancet. 1997 Jun 21;349(9068):1787-92. PMID 9269212
- [Background] Ruggenenti P, Perna A, Remuzzi G. ACE inhibitors to prevent end-stage renal disease: when to start and why possibly never to stop: a post hoc analysis of the REIN trial results. Ramipril Efficacy in Nephropathy. J Am Soc Nephrol. 2001 Dec;12(12):2832-2837. doi: 10.1681/ASN.V12122832. PMID 11729254
- [Background] Bakris GL, Agarwal R, Anker SD, Pitt B, Ruilope LM, Rossing P, Kolkhof P, Nowack C, Schloemer P, Joseph A, Filippatos G; FIDELIO-DKD Investigators. Effect of Finerenone on Chronic Kidney Disease Outcomes in Type 2 Diabetes. N Engl J Med. 2020 Dec 3;383(23):2219-2229. doi: 10.1056/NEJMoa2025845. Epub 2020 Oct 23. PMID 33264825
- [Background] Heerspink HJL, Stefansson BV, Correa-Rotter R, Chertow GM, Greene T, Hou FF, Mann JFE, McMurray JJV, Lindberg M, Rossing P, Sjostrom CD, Toto RD, Langkilde AM, Wheeler DC; DAPA-CKD Trial Committees and Investigators. Dapagliflozin in Patients with Chronic Kidney Disease. N Engl J Med. 2020 Oct 8;383(15):1436-1446. doi: 10.1056/NEJMoa2024816. Epub 2020 Sep 24. PMID 32970396
- [Background] The EMPA-KIDNEY Collaborative Group; Herrington WG, Staplin N, Wanner C, Green JB, Hauske SJ, Emberson JR, Preiss D, Judge P, Mayne KJ, Ng SYA, Sammons E, Zhu D, Hill M, Stevens W, Wallendszus K, Brenner S, Cheung AK, Liu ZH, Li J, Hooi LS, Liu W, Kadowaki T, Nangaku M, Levin A, Cherney D, Maggioni AP, Pontremoli R, Deo R, Goto S, Rossello X, Tuttle KR, Steubl D, Petrini M, Massey D, Eilbracht J, Brueckmann M, Landray MJ, Baigent C, Haynes R. Empagliflozin in Patients with Chronic Kidney Disease. N Engl J Med. 2023 Jan 12;388(2):117-127. doi: 10.1056/NEJMoa2204233. Epub 2022 Nov 4. PMID 36331190
- [Background] Okpechi IG, Bello AK, Ameh OI, Swanepoel CR. Integration of Care in Management of CKD in Resource-Limited Settings. Semin Nephrol. 2017 May;37(3):260-272. doi: 10.1016/j.semnephrol.2017.02.006. PMID 28532555
- [Background] World Health Organization. Strengthening Health Systems to Improve Health Outcomes. https://www.who.int/healthsystems/ strategy/en/. 2007. Accessed February 26, 2021
- [Background] Commission NP. The Malawi Noncommunicable Diseases & Injuries Poverty Commission Report. Lilongwe: Malawi Ministry of Health, 2018. http://www.ncdipoverty.org/malawi-report
- [Background] Crampin AC, Dube A, Mboma S, Price A, Chihana M, Jahn A, Baschieri A, Molesworth A, Mwaiyeghele E, Branson K, Floyd S, McGrath N, Fine PE, French N, Glynn JR, Zaba B. Profile: the Karonga Health and Demographic Surveillance System. Int J Epidemiol. 2012 Jun;41(3):676-85. doi: 10.1093/ije/dys088. Epub 2012 Jun 22. PMID 22729235